CLINICAL TRIAL: NCT04164602
Title: New Onset of DiabetEs in aSsociation With Pancreatic Cancer
Brief Title: The Occurence of Pancreatic Cancer Studied in Association With Newly Diagnosed Diabetes in the Elderly
Acronym: NODES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Collaborators: Hungarian Pancreatic Study Group (HPSG) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 41085-6/2019EÜIG
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus; Diabetes; Diabetes Mellitus, Type 2; Diabetes type2; Cancer of Pancreas; Pancreas Neoplasm; Pancreas Adenocarcinoma; Pancreatic Cancer
Keywords: new-onset diabetes mellitus; pancreatic cancer; biomarker; screening
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — C-peptide and glutamic acid decarboxylase antibodies (GADA) will be determined to classify diabetes CA 19-9 will be taken at every 12 months Blood to biobank will be taken at every 12 months. Biomarkers will be determined comparing metabolite levels in plasma samples from patients diagnosed with pancreatic cancer and diabetic cancer-free patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients with newly diagnosed diabetes: 1. Group with exposure: patients over 60 years of age with diabetes diagnosed within six months (newly diagnosed)
  2. Control Group: without exposure; patients over 60 years, without diabetes.

SUMMARY:
The aim of this study is to accomplish the early diagnosis of pancreatic cancer, in patients over 60 years of age with newly diagnosed diabetes. Only patients with type 2 diabetes are meant to be included. The early diagnosis of pancreatic cancer could be the way to enable efficient cure for the patients.

DETAILED DESCRIPTION:
The prognosis of pancreatic cancer is extremely unpleasant, which can be characterized with a 5-year survival rate of only about 6%. The disease usually pertaining no symptoms at the early phase, this might be one of the causes why it is discovered at a relatively late, inoperable stage - in most of the cases. The success of reducing the high mortality rate of pancreatic cancer could depend on the significant development of early diagnosis and also prevention programs. As the lifetime prevalence of pancreatic cancer is only 1.39%, screening through the whole population would be extremely expensive and difficult to manage. It would be recommended for all the individuals at high risk for pancreatic cancer to be examined. Patients newly diagnosed with diabetes have an approximately 8-fold risk for developing this type of cancer, compared to the average population. In addition to this age is also known as an independent risk factor for the pancreatic cancer. Recently there has been a biomarker panel identified, which may distinguish between pancreatic cancer and chronic pancreatitis in patients, with high sensitivity and specificity. The aim of this study is to accomplish the early diagnosis of pancreatic cancer, in patients over 60 years of age with newly diagnosed diabetes mellitus using a specific biomarker panel. Only patients with type 2 diabetes are meant to be included. Diabetes is classified by determining C-peptide levels, representing the endogenous insulin synthesis, also detecting glutamic acid decarboxylase (GADA) antibodies, the autoantibody against the pancreatic islet cells. The early diagnosis of pancreatic cancer could be the way to enable efficient cure for the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients over 60 years of age
* diabetes diagnosed within six months (newly diagnosed)
* signed written informed consent

Exclusion Criteria:

* continous alcohol abuse
* chronic pancreatitis
* previous pancreas operation/pancreatectomy
* pregnancy
* present malignant disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who meet the inclusion criteria will be included in the study at the participating centers at the Diabetology of the specialized outpatient clinics and also the GP practices involved.
  Patients, regardless of their gender as the daily patient population over 60 years of age and diagnosed with diabetes within 6 months.
Sampling Method: Probability Sample
Enrollment: 2522 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of pancreatic ductal adenocarcinoma in patients with new-onset diabetes | 36 months
  This will be evaluated using yes/no questions on carcinoma ductale, then the data will be summarized in order to determine the incidence.

SECONDARY OUTCOMES:
mortality of pancreatic ductal adenocarcinoma in new-onset diabetic patients | 36 months
  This will be evaluated using yes/no questions as part of a questionnaire filled out by the doctor who examines the patients.
the proportion of localised and resectable pancreatic ductal adenocarcinoma | 36 months
  Will be appraised after collecting and summarizing all the collected medical information.
change in body weight | 36 months
  Measuring the body weight of the patient and the data is recorded in the questionaire.
Change in fasting blood glucose and HbA1c | 36 months
  Based on the laboratory measurements.
Antidiabetic medications and the risk of pancreatic ductal adenocarcinoma | 36 months
  According to the anwers of the patients recorded on the questionnaire.
presence of concomitant diseases | 36 months
  According to the physical examinations and laboratory parameters also the anwers of the patients recorded on the questionnaire
smoking and alcohol intake | 36 months
  According to the anwers of the patients recorded on the questionnaire.
The sensitivity, specificity, positive and negative predictive values, and accuracy of the biomarker test | 36 months
  Will be appraised after collecting and summarizing all the collected medical information.
Cost-benefit analysis | 36 months
  Healthcare cost spent on each patient will be calculated by a healthcare economist after the trial is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Péter Hegyi, MD, PhD, DSc, Study Chair — Insitute for Translational Medicine, Medical School, University of Pécs, HU; László Czakó, MD, PhD, DSc, Principal Investigator — First Department of Medicine University of Szeged, HU
Locations (1):
- First Department of Medicine, Albert Szent-Györgyi Medical and Pharmaceutical Centre, University of Szeged, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rahib L, Smith BD, Aizenberg R, Rosenzweig AB, Fleshman JM, Matrisian LM. Projecting cancer incidence and deaths to 2030: the unexpected burden of thyroid, liver, and pancreas cancers in the United States. Cancer Res. 2014 Jun 1;74(11):2913-21. doi: 10.1158/0008-5472.CAN-14-0155. PMID 24840647
- [Result] Brand RE, Lerch MM, Rubinstein WS, Neoptolemos JP, Whitcomb DC, Hruban RH, Brentnall TA, Lynch HT, Canto MI; Participants of the Fourth International Symposium of Inherited Diseases of the Pancreas. Advances in counselling and surveillance of patients at risk for pancreatic cancer. Gut. 2007 Oct;56(10):1460-9. doi: 10.1136/gut.2006.108456. PMID 17872573
- [Result] Chari ST, Leibson CL, Rabe KG, Ransom J, de Andrade M, Petersen GM. Probability of pancreatic cancer following diabetes: a population-based study. Gastroenterology. 2005 Aug;129(2):504-11. doi: 10.1016/j.gastro.2005.05.007. PMID 16083707
- [Result] Huxley R, Ansary-Moghaddam A, Berrington de Gonzalez A, Barzi F, Woodward M. Type-II diabetes and pancreatic cancer: a meta-analysis of 36 studies. Br J Cancer. 2005 Jun 6;92(11):2076-83. doi: 10.1038/sj.bjc.6602619. PMID 15886696
- [Result] Ben Q, Xu M, Ning X, Liu J, Hong S, Huang W, Zhang H, Li Z. Diabetes mellitus and risk of pancreatic cancer: A meta-analysis of cohort studies. Eur J Cancer. 2011 Sep;47(13):1928-37. doi: 10.1016/j.ejca.2011.03.003. Epub 2011 Mar 31. PMID 21458985
- [Result] Pannala R, Basu A, Petersen GM, Chari ST. New-onset diabetes: a potential clue to the early diagnosis of pancreatic cancer. Lancet Oncol. 2009 Jan;10(1):88-95. doi: 10.1016/S1470-2045(08)70337-1. PMID 19111249
- [Result] Illes D, Terzin V, Holzinger G, Kosar K, Roka R, Zsori G, Abraham G, Czako L. New-onset type 2 diabetes mellitus--A high-risk group suitable for the screening of pancreatic cancer? Pancreatology. 2016 Mar-Apr;16(2):266-71. doi: 10.1016/j.pan.2015.12.005. Epub 2015 Dec 23. PMID 26777407
- [Result] Hart PA, Kamada P, Rabe KG, Srinivasan S, Basu A, Aggarwal G, Chari ST. Weight loss precedes cancer-specific symptoms in pancreatic cancer-associated diabetes mellitus. Pancreas. 2011 Jul;40(5):768-72. doi: 10.1097/MPA.0b013e318220816a. PMID 21654538
- [Result] Munigala S, Singh A, Gelrud A, Agarwal B. Predictors for Pancreatic Cancer Diagnosis Following New-Onset Diabetes Mellitus. Clin Transl Gastroenterol. 2015 Oct 22;6(10):e118. doi: 10.1038/ctg.2015.44. PMID 26492440
- [Result] Mayerle J, Kalthoff H, Reszka R, Kamlage B, Peter E, Schniewind B, Gonzalez Maldonado S, Pilarsky C, Heidecke CD, Schatz P, Distler M, Scheiber JA, Mahajan UM, Weiss FU, Grutzmann R, Lerch MM. Metabolic biomarker signature to differentiate pancreatic ductal adenocarcinoma from chronic pancreatitis. Gut. 2018 Jan;67(1):128-137. doi: 10.1136/gutjnl-2016-312432. Epub 2017 Jan 20. PMID 28108468
- [Derived] Illes D, Ivany E, Holzinger G, Kosar K, Adam MG, Kamlage B, Zsori G, Tajti M, Svebis MM, Horvath V, Olah I, Marta K, Vancsa S, Zadori N, Szentesi A, Czako B, Hegyi P, Czako L. New Onset of DiabetEs in aSsociation with pancreatic ductal adenocarcinoma (NODES Trial): protocol of a prospective, multicentre observational trial. BMJ Open. 2020 Nov 19;10(11):e037267. doi: 10.1136/bmjopen-2020-037267. PMID 33444177